CLINICAL TRIAL: NCT07333248
Title: Strengthening Community -to- Hospital Eye Care Pathways From Boko Eye Care Center in Rural Assam - From Referral to Treatment
Brief Title: Strengthening Community- to- Hospital Eye Care Pathways From Boko Eye Care Center in Rural Assam
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seva Canada Society (Other)
Collaborators: Pragyaan Sustainable Health Outcomes Foundation (Unknown); Sri Sankaradeva Nethralaya (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SSDN/IARC/46/2025-NOV/7
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Cataract; Refractive Errors
Keywords: Referral completion; Cataract surgery uptake; Patient navigation; Community engagement; Rural eye care; Surgical acceptance; Assam; LMIC
MeSH Terms: conditions — Cataract; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Referral and Engagement (Experimental): Referral tracking, patient navigation, community awareness tools, standardized counseling, transport and financial facilitation mechanisms
  Interventions: Other: Experimental: Integrated Referral and Engagement Model

INTERVENTIONS:
Other: Experimental: Integrated Referral and Engagement Model — Referral tracking, patient navigation, community awareness tools, standardized counseling, transport and financial facilitation mechanisms

SUMMARY:
This operational research project aims to strengthen continuity of eye care delivery between community screening and hospital-based treatment in rural Assam by redesigning referral pathways from the Boko Eye Care Center (ECC) to Sri Sankaradeva Nethralaya (SSDN) base hospital. Despite active outreach in the Boko region from the Boko ECC through conducting regular outreach screenings, less than 30 percent of patients referred to the base hospital actually arrive for evaluation and less than 25 percent of those advised for surgery proceed to treatment. The proposed study addresses these gaps by examining behavioural, structural and logistical barriers to referral completion and surgical uptake, and by implementing a coordinated patient-centered referral and engagement strategy.

The proposed intervention comprises of five sequential components: (1) root cause analysis to identify bottlenecks and facilitators in the current referral pathway, (2) community engagement activities to improve awareness and proactive health-seeking behaviour, (3) implementation of an integrated referral and engagement model supported by trained community team and structured referral tracking, (4) strengthening referral completion through patient navigation, scheduled transport and follow-up reminders, and (5) enhancement of surgical acceptance through standardized counseling, affordability support and social reinforcement. The outcomes will be measured prospectively, focusing on increase in hospital footfall from the Boko catchment area, proportion of referred patients who complete hospital visits, and proportion of patients who were advised for surgery and had undergone the procedure. The proposed project aims to achieve a minimum of 70 percent referral completion and 45 percent surgical conversion by the end of the 36-month study period.

DETAILED DESCRIPTION:
This 36-month prospective mixed-methods operational research project is designed to strengthen the referral-to-treatment continuum for rural eye care by improving patient flow from community screening activities at the Boko Eye Care Center (ECC) in Kamrup (Rural), Assam, to Sri Sankaradeva Nethralaya (SSDN) base hospital in Guwahati. Despite extensive outreach activities, the Boko ECC indicated comparatively weak conversion from community identification to hospital attendance and surgical uptake, with recent service statistics indicating less than 30 percent of referred patients reaching the base hospital and less than 25 percent undergoing advised surgery. The gap could be driven by a combination of behavioural barriers (fear, stigma, low motivation, skepticism about surgery), socioeconomic constraints (inability to pay, transport challenges, lost wages), logistical barriers (distance, lack of navigation or follow-up systems), and competition from private providers offering more proactive patient-handling systems. This study aims to systematically identify and address these barriers by developing and evaluating a context-sensitive, patient-centered model that would integrate community engagement, structured patient navigation, standardized counseling and financial facilitation.

The study will be conducted in three phases: a diagnostic research phase, an implementation phase and an evaluation phase. Phase 1 (Months 0-6) would include baseline referral pathway analysis and a root cause analysis using mixed methods. A quantitative baseline data will be extracted from screening registers, referral records and hospital information systems to determine referral uptake and surgical conversion. Qualitative data will be collected through in-depth interviews, focus group discussions, staff consultations and participatory group discussions with patients, family members, outreach field workers, and ECC service providers. The output of this phase will be a synthesized list of bottlenecks and facilitators that will guide intervention refinement.

Phase 2 (Months 7-18) would focus on community engagement and response building. A Community Engagement Toolkit (CET) will be developed and pretested for discussions in local settings and peer influences from successfully treated patients. The Community Eye Health workers and SSDN's dedicated ASECA workers will be trained to reinforce awareness and normalize hospital-based treatment. The engagement activities will be monitored using attendance logs, communication audit checklists and community feedback interviews. A midline survey will be conducted to capture changes in awareness, risk perception and care-seeking behaviour compared to baseline.

Phase 3 (Months 13-36) would focus on implementation of an integrated referral and engagement model informed by findings from Phase 1 and behaviour change momentum from Phase 2. This model would include structured referral tracking at the point of screening, scheduled referral appointments, active follow-up reminders, trained navigators to accompany patients, transport coordination to SSDN and standardized surgical counseling sessions at both the ECC and at the base hospital. The Counseling will follow a documented script that would address disease severity, outcome expectation, fear reduction, cost transparency and postoperative course. The field navigators will maintain referral completion forms and navigation logs. The fidelity of intervention delivery will be supervised through periodic observation and score-based assessment.

The outcome assessment will be done throughout implementation and formally at the end of the study. The primary outcome would be the referral completion rate (defined as the proportion of referred patients attending the SSDN base hospital within 90 days) and the proportionate change in hospital footfall from the Boko catchment area. The secondary outcome would include surgical conversion rate, defined as the percentage of patients advised for surgery who undergo the procedure within 90 days of referral. Trend analyses will also examine whether community engagement contributes to an increase in first-time eye screening attendance. Quantitative analysis will use descriptive statistics, chi-square tests for comparison of proportions, multivariate logistic regression to examine adjusted effects and interrupted time-series analysis to assess change in monthly conversion patterns. Qualitative transcripts will undergo thematic analysis, and the findings will be triangulated with quantitative results to understand mechanisms of change.

The proposed project has both scientific and public health relevance. Scientifically, the project would generate implementation evidence on strengthening referral systems in low-resource settings where passive referrals could lead to bottlenecks in treatment completion. Operationally, it would blend behavioural and structural interventions through toolkits, navigation systems and financial facilitation to reduce preventable blindness. The proposed project is fully aligned with WHO's Integrated People-Centered Eye Care framework and India's National Programme for Control of Blindness and Visual Impairment. Upon completion of the project, the findings are expected to demonstrate feasible and scalable approaches for optimizing patient referral and surgical acceptance in rural Assam, with potential to be adapted across SSDN's network of other 19 primary eye care centers. The expected outcomes include at least 70 percent referral completion, 45 percent surgical conversion and 30 percent rise in hospital footfall from the Boko ECC catchment by the end of 36 months. The broader aim is to establish a durable system of community-to-hospital linkage that would ensure timely access to sight-restoring care for underserved populations.

ELIGIBILITY:
Inclusion Criteria:

Adults diagnosed with eye conditions requiring referral or surgical treatment.

Exclusion Criteria:

Patients requiring emergency treatment, patients medically unfit for surgery, or patients unwilling to participate.

Eligibility: Enrolment criteria: Participants will be enrolled consecutively at the time of screening in community outreach camps and at the Boko Eye Care Center if they meet the following operational criteria:

i. Adult (≥18 years) with a diagnosed eye condition requiring referral to Sri Sankaradeva Nethralaya for tertiary evaluation or surgical treatment, as determined by the examining optometrist/ophthalmologist.

ii. Resident of the Boko Eye Care Center catchment area (villages linked to the Eye Care Center under Sri Sankaradeva Nethralaya outreach).

iii. Patients willing to provide informed consent to participate in the study and to allow follow-up for referral completion and surgical acceptance outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Referral completion rate to base hospital | 36 months
  Referral completion rate to base hospital

SECONDARY OUTCOMES:
Surgical conversion rate among patients advised for surgery | 36 months
  Surgical conversion rate among patients advised for surgery

OTHER OUTCOMES:
Increase in overall hospital footfall originating from Boko catchment area | 36 months
  Increase in overall hospital footfall originating from Boko catchment area

CONTACTS AND LOCATIONS:
Overall Officials: Priya Adisesha Reddy, Study Director — Seva Canada Society
Locations (1):
- Sri Sankaradeva Nethralaya, Guwahati, Assam, India

IPD SHARING:
Plan to Share IPD: No